CLINICAL TRIAL: NCT01850953
Title: Evaluating the Effects of Varenicline on Smoking Lapse in Smokers With and Without Schizophrenia: Implications for Treatment
Brief Title: Effects of Varenicline on Smoking Lapse in Smokers With and Without Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Tony George, Clinical Directot, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 225/2012; GRAND 2012 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2013-05-06; First posted 2013-05-10 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Craving; Smoking; Schizophrenia
Keywords: Varenicline; Schizophrenia; smoking; Lapse
MeSH Terms: conditions — Smoking; Schizophrenia | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Placebo Comparator): This is a sugar pill that will be used as a placebo comparator.
  Interventions: Drug: Placebo
- Varenicline (Active Comparator): Varenicline will be titrated to steady-state levels of 2mg/day over 4 days (0.5mg BID for day 1 and 1.0mg BID for days 2-4) before testing at 2mg/day on days 5 and 6.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — This is an approved smoking cessation medication.
  Other Names: Champix, Chantix
  Arms: Varenicline
Drug: Placebo
  Arms: Sugar Pill

SUMMARY:
The objective of this study is to determine the mechanisms by which varenicline, an effective smoking cessation treatment, protects against relapse. Varenicline will be administered in smokers with schizophrenia and control smokers using a randomized, double-blind, cross-over design. Smokers will be asked to stop smoking overnight; the next day the ability to resist smoking will be assessed in a laboratory smoking lapse paradigm. Measures of tobacco craving, reinforcement and withdrawal-related cognitive dysfunction will be correlated with time to lapse. The results could have significant clinical implications by identifying mechanisms by which smokers with schizophrenia are at more risk for relapse than the general population, leading to the development of more effective smoking cessation therapies.

DETAILED DESCRIPTION:
One way to facilitate medication development for smoking cessation is through the use of human laboratory paradigms that can provide an efficient, cost-effective and mechanistic evaluation of a medication signal on smoking behavior and bridge pre-clinical studies and costly clinical trials. This study will take advantage of the recent development and validation of a smoking lapse procedure to evaluate the effects of varenicline in smokers with and without schizophrenia. We will extend our recent work with varenicline by relating its effects on reinforcement, craving and cognition to clinical outcome (i.e., lapse - a strong predictor of relapse). It is pertinent to study smokers with schizophrenia because as smoking rates decline in the general population we will be left with a group of'hardcore' smokers for whom current smoking cessation strategies have limited efficacy.

The objective of this study is to determine the effect of varenicline versus placebo, on time to lapse, as a function of craving, reinforcement and cognitive dysfunction, in smokers with and without schizophrenia. We hypothesize that:

1. Smokers with schizophrenia will have reduced ability to resist smoking during the placebo condition compared to controls; and secondarily, this will be related to the higher levels of cognitive dysfunction during abstinence.
2. Varenicline will increase the ability to resist smoking in both control and schizophrenia smokers; and secondarily, this will be mediated via its effects on cognition in smokers with schizophrenia, and its effects on craving in control smokers.

The exploratory aims are to determine:

1. Varenicline's effect on cue-reactivity in smokers with and without schizophrenia and its relationship to time to lapse.
2. Varenicline's effects on tobacco reinforcement and its relationship to ad lib smoking in the lapse period

The current study will advance the development of tobacco addiction treatments in the following ways: 1) Identification of mechanisms by which varenicline facilitates abstinence in different subtypes of smokers (schizophrenia vs. controls) is critical to improve treatment response. 2) Identification of predictors of relapse in different subtypes of smokers (schizophrenia vs. controls) could guide future medication development efforts. 3) Relating measures of tobacco abstinence and addiction collected in the laboratory to proxy measures of treatment outcome (i.e., smoking lapse) will provide further validation that evaluation of medications in such paradigms is a useful and cost-effective screening strategy. 4) Our approach could also be used to identify smokers most at risk for tobacco abstinence symptoms who would benefit from treatments targeting the most prominent aspects of withdrawal. This could lead to improved health outcomes in smokers.

ELIGIBILITY:
Inclusion Criteria:

* Cigarette Smokers (smoke ≥ 10 cigarettes per day)
* non-treatment seeking (i.e., not trying to quit as indicated by <7 on the contemplation ladder)
* aged 18-55
* Intelligence Quotient (IQ) ≥80 on the Wechsler Test of Adult Reading [89]
* Fagerstrom Test of Nicotine Dependence (FTND) ≥4 [90]
* Patients must meet Structured Clinical Interview for the diagnostic and Statistical Manual for Mental Disorders (SCID-IV) diagnosis criteria for schizophrenia or schizoaffective disorder; be in stable remission from positive symptoms of psychosis as judged by a Positive and Negative Syndrome Scale (PANSS) positive score total score <70, and receiving a stable dose of antipsychotics for >1month.
* Control participants will not be taking any psychotropic medications at the time of enrollment and will not meet diagnostic criteria for any Axis I disorder, except past history of major depression or an anxiety disorder if in remission for at least one year.

Exclusion Criteria:

* substance use (except nicotine or caffeine) in the last month
* a history of alcohol/drug abuse in the 3 months before study enrollment
* use of opioids (meperidine, oxycodone, methadone, etc)
* current use of smoking cessation aids (e.g., nicotine replacement therapy, bupropion or varenicline
* pregnancy or nursing
* a history of renal insufficiency or a hypersensitivity to varenicline (Champix®)
* a history of neurological illness like epilepsy or medical condition known to significantly influence neurocognitive function
* any other medical condition deemed relevant by the Qualified Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Time to Lapse | Day 6 of week 1 and week 2
  The objective of this study is to determine the effect of varenicline versus placebo, on time to lapse using a lapse paradigm.

SECONDARY OUTCOMES:
Cognitive Function | Day 6 of week 1 and week 2
  The secondary objectives of this study are to determine the effect of varenicline versus placebo, on time to lapse, as a function of craving, reinforcement and cognitive dysfunction, in smokers with and without schizophrenia
Tobacco craving | Day 6 of week 1 and week 2
  The secondary objectives of this study are to determine the effect of varenicline versus placebo, on time to lapse, as a function of craving, reinforcement and cognitive dysfunction, in smokers with and without schizophrenia
Tobacco withdrawal | Day 6 of week 1 and week 2
  The secondary objectives of this study are to determine the effect of varenicline versus placebo, on time to lapse, as a function of craving, reinforcement and cognitive dysfunction, in smokers with and without schizophrenia
Tobacco Reinforcement | Day 6 of week 1 and week 2
  The secondary objectives of this study are to determine the effect of varenicline versus placebo, on time to lapse, as a function of craving, reinforcement and cognitive dysfunction, in smokers with and without schizophrenia

CONTACTS AND LOCATIONS:
Overall Officials: Tony George, M.D., Study Director — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research